CLINICAL TRIAL: NCT05796492
Title: Fieldable Ultrasound Treatment to Enhance Inflammatory-Proliferative Phase Transition and Reduce Wound Healing Time
Brief Title: Ultrasound Treatment on Wound Healing Time
Acronym: GE-MTEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment/ enrollment issues
Sponsor: General Electric Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-22-00019
Record Dates: First submitted 2022-08-22; First posted 2023-04-03 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Burn Wound; 2nd Degree Burn of the Skin
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LOGIQ E10 Sham (Sham Comparator): The sham condition will consist of the ultrasound probe placed over the spleen with no energy applied.
  Interventions: Device: Ultrasound probe (no energy applied)
- LOGIQ E10 ultrasound Active (Active Comparator): The intervention condition will receive 10 minutes of splenic ultrasound daily.
  Interventions: Device: Pulsed splenic ultrasound

INTERVENTIONS:
Device: Pulsed splenic ultrasound — A General Electric LOGIQ E10 ultrasound machine with a C1-6-XD clear probe, will be used to selectively deliver pulsed ultrasound to the spleen.
  Other Names: Active ultrasound
  Arms: LOGIQ E10 ultrasound Active
Device: Ultrasound probe (no energy applied) — A General Electric LOGIQ E10 ultrasound probe will be placed over the spleen with no energy applied
  Arms: LOGIQ E10 Sham

SUMMARY:
This is a randomized, sham-controlled pilot study that will assess the safety and feasibility of splenic focused pulsed ultrasound treatment on burn wound healing time in 24 subjects (12 active ultrasound and 12 sham controls).

DETAILED DESCRIPTION:
The Central Hypothesis underlying this study is that splenic ultrasound stimulation activates the splenic anti-inflammatory pathway, thereby producing reduction in circulating macrophage cytokine production, reduction of neutrophil invasiveness, or induction of phenotypic transition in circulating immune cells (e.g., M1 to M2 transition in macrophages) in patients with partial thickness wounds that cover <20% body surface area.

Approximately 24 subjects will participate in this study. Male and female subjects of all races and ethnicities will be recruited for study from the ethnically diverse patient population of the LAC+USC Burn Center from the surrounding area.

Phase 0

Burn wound subjects will be screened and enrolled at the LAC+USC Burn Center located in Los Angeles, California. No other sites, neither regional nor outside of the United States are going to participate in enrollment of subjects.

A General Electric LOGIQ E10 ultrasound machine with a C1-6-XD clear probe, will be used to selectively deliver pulsed ultrasound to the spleen.

12 months.

28 days or until healed (whichever comes first)

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18 or older
* Second-degree burn wounds of less than 20% total body surface area (TBSA)
* No active wound infection at screening based on clinical criteria
* Able to provide written informed consent

Exclusion Criteria:

* Wounds determined by study clinicians to be ineligible, including those that may inhibit access to the spleen for the ultrasound procedure
* Participating in another research study that may affect the conduct of results of this study
* BMI > 30
* Having or exhibiting any of the following:

  * Previous surgery of the spleen, esophagus, stomach, duodenum, or liver, including splenectomy
  * End stage renal disease and/or uremia
  * Active malignancy
  * Previous leukemia and/or lymphoma
  * Human immunodeficiency virus infection or AIDS
  * Rheumatoid arthritis or other immune-mediated diseases (e.g., inflammatory bowel disease
  * Arrythmias, including but not limited to, atrial fibrillation, atrial flutter, clinically significant bradycardia, ventricular arrhythmias, and A-V block
  * Implanted pacemaker or cardioverter/debribrillator
  * History of unstable angina, angioplasty or coronary arterial by-pass grafting surgery
  * History of stroke or TIA
  * Untreated thrombosis or bleeding disorders
  * Currently implanted vagus nerve stimulator
  * Currently implanted spinal cord stimulator or other chronically implanted electronic device
* Receiving oral, topical, rectal, or parenteral corticosteroids in an unstable dose 4 weeks prior to baseline visit
* Any immunosuppressive or cytotoxic medications
* Clinically relevant history of alcohol or drug abuse as determined by the investigator including:

  * alcohol consumption within 4 days of the baseline visit
  * tobacco or nicotine product use within the past 1 month
  * recreational drug use within the past 1 month
* Pregnant or breast feeding
* Unable or unwilling to comply with study procedures
* Have recently (within 3 months) been diagnosed with COVID, or have ever been diagnosed with long COVID
* Have an autoimmune disorder, such as, rheumatoid arthritis or lupus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse device effects (ADEs) | Days 1 -28
  Review of anticipated device effects after splenic ultrasound insonification in subjects with partial thickness wounds that cover <20% body surface area.
Median time to re-epithelialization using advanced digital imaging | 28 days or until healed (whichever comes first)
  Re-epithelialization measured by digital planimetry

SECONDARY OUTCOMES:
Difference in groups in pain measured visual analog scale, (VAS) | Days 7, 14, 21 and 28
  Pain, scale 0-10 with 10 being worst outcome
Difference in groups in itch measured visual analog scale, (VAS) | Days 7, 14, 21 and 28
  Itch, scale 0-10 with 10 being worst outcome
Difference in groups in non-invasive perfusion measured visual analog scale, (VAS) | Days 7, 14, 21 and 28
  Doppler perfusion, scale 0-10 with 10 being worst outcome
Referral to scar management specialist | Days 7, 14, 21 and 28
  Scar management
Scar assessments using Patient and Observer Scar Assessment Scale (POSAS) | Days 7, 14, 21 and 28
  A 5 point score ranging from 1 (normal pigmentation, no itching) to 5 (worst imaginable scar or sensation).
Multiplexed analysis of plasma levels of inflammatory cytokines | Days 7, 14, 21 and 28
  Plasma levels of inflammatory cytokines, lab range values
Flow cytometry analysis of phenotype of macrophage, neutrophil, and T lymphocyte populations | Days 7, 14, 21 and 28
  Phenotype of macrophage, neutrophil, and T lymphocyte, lab range values

CONTACTS AND LOCATIONS:
Overall Officials: David Armstrong, DPM, MD, PhD, Principal Investigator — USC Limb Preservation Consortium
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States